CLINICAL TRIAL: NCT00357474
Title: A Multicenter, Randomized, Controlled Trial of the Effective Therapy for Multiple, Small Hepatocellular Carcinomas: Comparing Transarterial Chemoembolization With Percutaneous Ethanol Injection Therapy.
Brief Title: Comparison Study of Transarterial Chemoembolization and Percutaneous Ethanol Injection for Multiple, Small HCCs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jung-Hwan Yoon, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 07-2006-010
Record Dates: First submitted 2006-07-26; First posted 2006-07-27 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Hepatocellular Carcinoma
Keywords: HCC, TACE, PEIT
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- chemotherapy (Active Comparator): Transarterial chemoembolization (TACE)
  Interventions: Procedure: Transarterial chemoembolization
- ethanol (Active Comparator): Percutaneous ethanol injection therapy (PEIT)
  Interventions: Procedure: Percutaneous ethanol injection therapy

INTERVENTIONS:
Procedure: Transarterial chemoembolization — lipiodol, adriamycin and/or mitomycin
  Other Names: TACE
  Arms: chemotherapy
Procedure: Percutaneous ethanol injection therapy — 99% ethanol 2-4cc per one session, two to three sessions per single procedure for one week
  Other Names: PEIT
  Arms: ethanol

SUMMARY:
The purpose of this study is to choose the preferred treatment modality for multiple, small hepatocellular carcinomas.

DETAILED DESCRIPTION:
To compare the below things between PEIT group and TACE group

1. Survival

   1. 5 year overall survival rate
   2. Disease free survival rate
2. Recurrence a. recurrence rate

ELIGIBILITY:
Inclusion Criteria:

* The evidences of HBV(+) &/or HCV(+) infection or liver cirrhosis
* Two to three tumor nodules with Child-Pugh classification A or single to three tumor nodules with Child-Pugh classification B
* The maximal, longest diameter of tumor mass measured by CT finding should be less than 2 cm.
* 1) Only for newly detected HCCs which were not treated before or 2) If treated before, it should be noted that there is no evidence of recurrence within the latest 6 months and, and also it should be remotely recurred more than 2cm apart from primary lesion.
* It should be compatible with the typical findings of HCCs radiologically(MD CT or dynamic MRI)

Exclusion Criteria:

* In case of hepatic vein or portal vein invasion radiologically(CT or MRI)

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2005-10; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
overall survival rate | 5 year

SECONDARY OUTCOMES:
Disease free survival rate and recurrence rate | 5 year

CONTACTS AND LOCATIONS:
Overall Officials: J H Yoon, Professor, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul NUH, Seoul, Chongno-gu, South Korea